CLINICAL TRIAL: NCT00055848
Title: Familial Factors in the Development of Colon Cancer
Brief Title: Genetic Study of Familial Factors in Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150008; CALGB-150008; CDR0000271314 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Cytogenetic Analysis; Chromosome Mapping; Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients donate blood samples for analysis of colorectal susceptibility genes. Patients also complete a questionnaire regarding family cancer history.
  A certificate of confidentiality protecting the identity of research participants in this project has been issued by the National Cancer Institute.
  Participants do not receive the results of the genetic testing, and the results do not influence the type or duration of treatment.
  Interventions: Genetic: cytogenetic analysis; Genetic: gene mapping; Genetic: microarray analysis

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: gene mapping
Genetic: microarray analysis

SUMMARY:
RATIONALE: Genetic studies may help in understanding the genetic processes involved in the development of some types of cancer.

PURPOSE: Clinical trial to study the cancer-related genes in patients who have colon cancer or adenomatous polyps.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify human colon neoplasia susceptibility genes in patients with colon cancer or adenomatous polyps.
* Correlate the inheritance of novel susceptibility alleles for adenomatous polyposis of the colon with colon neoplasia in these patients.
* Correlate colon neoplasia susceptibility with the presence of COX-2, sPLA2, and DNMT genes in these patients.
* Identify a novel gene that governs increased susceptibility to colon adenoma and cancer in the genome of these patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer or polyps at age 70 or under
* Has a living full sibling with diagnosis of colon cancer or polyps at age 70 or under
* No history of familial adenomatous polyposis syndrome
* No hereditary nonpolyposis colon cancer, according to Amsterdam criteria
* No known I1370K adenomatous polyposis of the colon susceptibility variant
* Enrolled on 1 of the following clinical trials:

  * CLB-9581
  * CLB-89803
  * CLB-80001 NOTE: Patients do not need to be receiving protocol therapy. Patients who are outside the treatment protocol's follow-up range are eligible. Patients who discontinued therapy for any reason, including toxic effects, are eligible.

PATIENT CHARACTERISTICS:

Age

* 70 and under at diagnosis

Other

* No significant psychiatric illness that would preclude giving informed consent
* No inflammatory bowel disease (in patient or sibling)

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with colon cancer or polyps age 70 or under. Specifically, patients previously enrolled on CLB-9581, CLB-89803 and CLB-80001.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2001-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica M. Bertagnolli, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina, United States